CLINICAL TRIAL: NCT00800059
Title: A Dose Escalation Study of Total Marrow Irradiation (TMI) and Autologous Stem Cell Transplantation (ASCT) for the Treatment of Relapsed or Refractory Multiple Myeloma (MM)
Brief Title: Total Marrow Irradiation & Autologous Stem Cell Transplantation for Relapsed or Refractory Myeloma
Acronym: TMI-ASCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008519-01H
Record Dates: First submitted 2008-11-27; First posted 2008-12-01 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma
Keywords: Relapse; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment with TMI and autologous Stem Cell transplant
  Interventions: Radiation: Total Marrow Irradiation

INTERVENTIONS:
Radiation: Total Marrow Irradiation — Total Marrow Irradiation delivered by chemotherapy delivered to cohorts of patients in a dose escalation. The initial cohort will receive 14 Gy. If tolerated subsequent cohorts will receive an additional 2 Gy until the maximum tolerated dose or 28 Gy is reached.
  Other Names: TMI

SUMMARY:
The investigators hypothesize that conformal radiation will allow the administration of higher doses of external beam radiation to marrow based malignancies than total body irradiation (TBI)without increasing the toxicity to normal tissues beyond that induced by TBI. Further,the investigators hypothesize that this will result in an improvement in disease response and disease control for patients with multiple myeloma. This is a dose escalation study of TMI with the primary objective of determining the maximum tolerated dose of TMI when followed by aHSCT in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet all of the following criteria to be eligible for the study. These will be evaluated within the four weeks prior to enrolment.
* Subject must have primary refractory or relapsed multiple myeloma.
* Subject must have a measurable serum or urine monoclonal gammopathy at the time of their latest relapse.
* Subject must meet institutional guidelines for autologous HSCT with adequate renal, cardiac, pulmonary and hepatic function.
* An autologous hematopoietic stem cell graft containing more than 2.5 x 106 CD34+ cells/kg must be cryopreserved and available for transplantation.
* Subject must be of age more than 18 and less than 60 years.
* Subject must have an ECOG performance score of 0,1, or 2.
* Subject must have the ability to comply with the protocol visit schedule and other protocol requirements.

Exclusion Criteria:

* A subject meeting any of the following criteria is not eligible for participation in the study:
* Subject with non-secretory multiple myeloma or any plasma cell disorders other that MM.
* Subjects that have not received previous therapy with adequate intense corticosteroids for multiple myeloma.
* Subjects with a severely limited life expectancy by concomitant illness, defined as a life-expectancy of less than 6 months.
* Subjects who have previously received radiation treatments or other neoplastic disorders.
* Subjects with a history of non-compliance in other studies.
* Pregnant or lactating female subjects.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2008-11; Primary Completion 2020-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of TMI when followed by aHSCT in patients with relapsed or refractory multiple myeloma | 30 days from the time of aSCT

SECONDARY OUTCOMES:
The frequency and timing of engraftment following TMI and aHSCT | within 30 days of aHSCT
The early morbidity and mortality associated with TMI and aHSCT | 30 days from aHSCT
The intermediate morbidity and mortality associated with TMI and aHSCT | 100 days from aHSCT
The late morbidity of TMI | Beyond 6 months after transplantaton

CONTACTS AND LOCATIONS:
Overall Officials: Harold L Atkins, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada